CLINICAL TRIAL: NCT04104243
Title: Power-Up: An Effectiveness Trial of the Diabetes Prevention Program Tailored for Men
Brief Title: Power-Up: An Effectiveness Trial of the Diabetes Prevention Program
Acronym: Power-Up
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: New York City Department of Health and Mental Hygiene (Other Government); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2019-10343; 5R01DK121896-04 (NIH); 2019-10343 (Other: Einstein - IRB ID)
Record Dates: First submitted 2019-09-19; First posted 2019-09-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Type 2 Diabetes; Pre-Diabetes
Keywords: Pre-Diabetes; Men's Health; Type 2 Diabetes; Racial Disparities
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance

STUDY DESIGN:
Intervention Model Description: There will be 6 intervention cycles. Approximately 50 men will be randomized 1:1 to each study arm. There will be 4 control cycles for every intervention workshop. Therefore we will have 6 intervention workshops and 24 control workshops. The participants will be randomized to either undergo Power-Up or standard Diabetes Prevention Program sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Power-Up (Experimental): Participants randomized to this arm will undergo 16 classes tailored for men, that discuss food choices, physical activity, and managing stress over 6 months, which are called the core, and 6 classes over the following 6 months, which is called the maintenance phase.
  Interventions: Other: Men-Tailored DPP (Power-Up)
- Standard NDPP (National Diabetes Prevention Program) (No Intervention): Participants randomized to this arm will undergo 16 mixed gender classes that discuss food choices, physical activity, and managing stress over 6 months which are called the core and 6 classes over the following 6 months which is called the maintenance phase.

INTERVENTIONS:
Other: Men-Tailored DPP (Power-Up) — Evaluating whether a diabetes prevention program (DPP) tailored for men (Power-Up) will show better or similar percent weight loss and retention than a standard mixed-gender DPP
  Arms: Power-Up

SUMMARY:
The goal of this study is to address the risk of diabetes among men by creating a Diabetes Prevention Program (DPP) tailored to men.

DETAILED DESCRIPTION:
The rising epidemic of type 2 diabetes is a major cause of disability and death that disproportionately affects men. Compared to women, men have much worse health and higher death rates for several chronic conditions, including diabetes. The National Diabetes Prevention Program (NDPP) has been shown to help decrease the chances of developing type 2 diabetes. The NDPP has shown the value of lifestyle change for weight loss and diabetes prevention. The Power-Up study is being done because although the evidence points to the effectiveness of the Diabetes Prevention Program (DPP), men are less likely to be engaged or participate in DPP.

The Power-up study was designed to see whether a DPP tailored for men can help improve engagement, participation, and results for men. Participants will be randomized to either undergo the Power-Up or standard NDPP classes. An assessment of whether a DPP created for men will increase participation in the program and decrease the risk for diabetes as compared to the standard NDPP. Power-Up is designed to Aim 1) Assess the effect of Power-Up vs. standard care NDPP on percent weight loss among men at risk for diabetes; Aim 2) Compare engagement of minority men at risk for diabetes in Power-Up vs. standard care NDPP; and Aim 3) Evaluate the Reach, Effectiveness, Adoption, Implementation, and Costs of Power-Up using the RE-AIM framework. The Power-Up intervention is tailored to the needs and preferences of men and uses: a) men coaches; b) men-only groups; c) messaging tailored to be appreciated and motivational to men; d) adapted content that highlights issues relevant to men.

There are 22-28 classes over the course of 12 months for both Power-Up and standard NDPP. The classes are split into two phases which are called the core and the maintenance phases. The core phase of the program will consist of at least 16 classes over the first 6 months. After the core, participants will attend maintenance classes over the next 6 months. Participants will be asked over the course of the 12 months to complete surveys at three different times before, during, and after completing the classes.

The hypothesis is that men randomized to Power-Up will achieve significantly greater weight loss (% weight loss from baseline) at 16 weeks and 1 year than men randomized to the standard care, mixed-gender NDPP group (Aim 1). Evaluation of engagement and retention for Aim 2 is based on attendance records for Power-Up and NDPP sessions electronically collected by trained coaches and monitored by study staff. The standards will be followed for NDPP evaluation where engagement is defined as equal or greater than 4 core sessions attended and retention is defined as equal or greater than 9 sessions attended. There will be a collection of quantitative and qualitative data that will be rigorously evaluated: the reach of our recruitment, broader patient-important indicators of effectiveness, adoption at the practice level, and implementation of the intervention (Aim 3).

Enrollment consists of 300 participants through our health system partners. Men will be randomized 1:1 to either the Power-Up intervention arm or referred to the standard NDPP at their clinic site. Consistent with current Centers for Disease Control and Prevention (CDC) standards and current NDPP practices of our health system partners, telephone make-up sessions will be offered by coaches in both conditions to men who miss in-person sessions.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Most recent HbA1c: 5.7%-6.4% (within last year) or Diabetes Risk Score >= 5
* Most recent BMI ≥ 25 (within last 6 months)
* Access to a device that can join sessions virtually either through a virtual conferencing application
* Have valid address and telephone contact information
* Have no plans to change their health system/primary care provider or move from their current, NYC area, address in the next year

Exclusion Criteria:

* Not physically able or willing to attend virtual, group-based sessions
* Unable to provide informed consent by telephone
* Unable or unwilling to complete baseline telephone surveys or follow-up surveys in English or Spanish

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — We are only enrolling men.
Enrollment: 301 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
Percent Weight Loss through 16 sessions | Up to 6 months, after the delivery of the 16th session (end of the core phase)
  Compare Percent Weight Loss through 16 sessions.
Percent Weight Loss through the 12 month trial | 12 Months (At end of maintenance phase)
  Compare Percent Weight Loss through the 12 month trial.

SECONDARY OUTCOMES:
Comparison of Engagement and Retention of Men vs Standard Diabetes Prevention Program | Up to 6 months, after the delivery of the 16th session (end of the core phase)
  Compare engagement of men at risk for diabetes in Power-Up vs. Standard DPP. The number of sessions scheduled.
Comparison of Engagement and Retention of Men vs Standard Diabetes Prevention Program | 12 Months (At end of the maintenance phase)
  Compare engagement of men at risk for diabetes in Power-Up vs. Standard DPP. The number of sessions attended. Engagement rates are characterized as attending at least 4 sessions. Retention is defined as attending 9 or more sessions. We expect men randomized to the Power-Up sessions will have greater engagement and retention rates than men randomized to standard care and referred to mixed-gender NDPP classes.

CONTACTS AND LOCATIONS:
Overall Officials: Earle Chambers, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Realmuto L, Kamler A, Weiss L, Gary-Webb TL, Hodge ME, Pagan JA, Walker EA. Power Up for Health-Participants' Perspectives on an Adaptation of the National Diabetes Prevention Program to Engage Men. Am J Mens Health. 2018 Jul;12(4):981-988. doi: 10.1177/1557988318758786. Epub 2018 Mar 15. PMID 29540130
- [Background] Walker EA, Weiss L, Gary-Webb TL, Realmuto L, Kamler A, Ravenell J, Tejeda C, Lukin J, Schechter CB. Power Up for Health: Pilot Study Outcomes of a Diabetes Prevention Program for Men from Disadvantaged Neighborhoods. Am J Mens Health. 2018 Jul;12(4):989-997. doi: 10.1177/1557988318758787. Epub 2018 Mar 15. PMID 29540129
- [Background] Gary-Webb TL, Walker EA, Realmuto L, Kamler A, Lukin J, Tyson W, Carrasquillo O, Weiss L. Translation of the National Diabetes Prevention Program to Engage Men in Disadvantaged Neighborhoods in New York City: A Description of Power Up for Health. Am J Mens Health. 2018 Jul;12(4):998-1006. doi: 10.1177/1557988318758788. Epub 2018 Mar 15. PMID 29540131
- [Derived] Chambers EC, Walker EA, Schechter C, Gil E, Herbert T, Diaz K, Gonzalez J. Virtual Diabetes Prevention Program Tailored to Increase Participation of Black and Latino Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jun 24;14:e64405. doi: 10.2196/64405. PMID 40554781

DOCUMENTS (1):
  • Informed Consent Form (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/43/NCT04104243/ICF_000.pdf